CLINICAL TRIAL: NCT05692167
Title: Dexmedetomidine as an Additive to Topical Versus Peribulbar Anesthesia for Cataract Surgery
Brief Title: Dexmedetomidine in Topical Versus Peribulbar Anesthesia for Cataract Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Lecturer of Anaesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Kafrelsheikh University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKSU 50-11-3
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Dexmedetomidine; Cataract Surgery; Peribulbar; Anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical dexmedetomidine group (Active Comparator): Patients will receive mixture of one milliliter of dexmedetomidine-HCl and local anesthetic
  Interventions: Drug: Topical dexmedetomidine
- Reginal dexmedetomidine group (Active Comparator): Patients will receive mixture of bupivacaine 0.5% (4.5 ml) + lidocaine 2% (4.5 ml) + dexmedetomidine 50 μg (1 ml) in peribulbar block
  Interventions: Drug: Reginal dexmedetomidine

INTERVENTIONS:
Drug: Topical dexmedetomidine — Patients will receive mixture of one milliliter of dexmedetomidine-HCl and local anesthetic
  Arms: Topical dexmedetomidine group
Drug: Reginal dexmedetomidine — Patients will receive mixture of bupivacaine 0.5% (4.5 ml) + lidocaine 2% (4.5 ml) + dexmedetomidine 50 μg (1 ml) in peribulbar block
  Arms: Reginal dexmedetomidine group

SUMMARY:
The aim of this study is to compare efficacy of dexmedetomidine as an additive to topical versus peribulbar anesthesia for cataract surgery

DETAILED DESCRIPTION:
Ocular surgery may be performed under topical, regional, or general anesthesia. The first recorded use of regional anesthesia for surgery was the instillation of cocaine into the conjunctival sac in 1884 by an Austrian ophthalmologist.

Davis and Mandel in 1986 described the peribulbar block, peribulbar block has delayed onset and need a higher volume of local anesthetic (LA) than a retrobulbar block. But the peribulbar block is away from intra-conal space and so produce fewer complication.

Dexmedetomidine is used as adjuvant to LA drugs in peripheral nerve block, brachial plexus block and intrathecal anesthesia with satisfactory results. A more recent study using dexmedetomidine (50 μg) with the peribulbar block before cataract surgery demonstrated an IOP decrease similar to IV dexmedetomidine administration and greater than a peribulbar block without dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification I or II who scheduled for eye surgery

Exclusion Criteria:

* Patients who are younger than 18 years
* The usual contraindications for regional anesthesia such as patients refusing LA
* Clotting abnormalities
* Impaired mental status
* Allergy to any of the study medications
* patients had the severe cardiac disease
* chronic obstructive lung disease and a history of sleep apnea
* contraindications to the use of dexmedetomidine
* history or significant cardiovascular disease risk factors
* significant coronary artery disease or any known genetic predisposition
* history of any kind of drug allergy
* drug abuse
* psychological or other emotional problems
* special diet or lifestyle
* clinically significant abnormal findings in physical examination
* electrocardiographic (ECG) or laboratory screening
* known systemic disease requiring the use of anticoagulants.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Inadvertent eye movement | 2 hours postoperatively
  Asses intra-ocular pressure (IOP) before injection of baseline and after a complete akinesia of the globe before surgical incision.

SECONDARY OUTCOMES:
Anesthesia-related complications | 2 hours postoperatively
  The patients will be asked whether the cataract surgery was more or less painful than having the needle used for intravenous infusions inserted into the back of the hand.
Sedation level | 2 hours postoperatively
  Numeric Rating Scale will be applied to grade the pain where 0 = no pain and 10 = extreme pain.
pain during and after the surgery | 2 hours postoperatively
  Immediately after surgery, patients will be asked to grade the pain felt during the operation, including the pain felt after delivery of topical or peribulbar anaesthesia.
Need for additional anesthesia during surgery and surgeon | During surgery
  The dose of additional needed anesthesia (fentanyl 0.5 µg/kg) during surgery will be recorded
Intraoperative difficulties | 2 hours postoperatively
  The surgeon will also be requested to grade any difficulties encountered during surgery immediately after the operation, using a 4-point scale, where 1 = no difficulty and 4 = extremely difficult

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed F Algyar, MD, Principal Investigator — Lecturer of Anaesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Kafrelsheikh University
Locations (1):
- Mohammed Fouad Mohamed Algyar, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available under a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after the end of the study